CLINICAL TRIAL: NCT01367197
Title: Randomised Study of the Effect of Exercise Training on Patients in Atrial Fibrillation
Brief Title: Study of the Effect of Exercise Training on Patients in Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Hvidovre University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Philip Osbak, MD, Hvidovre Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22300240
Record Dates: First submitted 2011-06-01; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Atrial Fibrillation
Keywords: exercise training; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention (No Intervention): Observation only
- Exercise training group (Experimental): Group exercise training, three times weekly high-intensity
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training — group based exercise training
  Arms: Exercise training group

SUMMARY:
PURPOSE Physical exercise is beneficial for patients with ischemic heart disease and chronic heart failure, while little is known about the effect in atrial fibrillation (AF). The investigators studied the effect of physical exercise on cardiac output (CO), max. exercise capacity, biomarkers and quality of life (Qol) in patients with AF in a randomised study of physical exercise training three times weekly for twelve weeks.

HYPOTHESIS Exercise training improves cardiac output (CO), max. exercise capacity, biomarkers and quality of life (Qol) in patients with AF.

METHODS Assessment of exercise capacity, CO, Qol, body composition, six minute walk test and muscular strength was performed before and after 12 weeks.

Resting echocardiography was done at baseline. CO was measured using impedance cardiography at rest and during maximal exercise testing on an ergometer bicycle. Body composition, muscular strength and six minutes walking capacity were measured before and after the training period. Qol was evaluated by the use of the standardized validated questionnaires Short Form 36 (SF-36) and the Minnesota Living with Heart Failure Questionnaire (MLHF-Q).

Training consisted of aerobic exercise at 70 percent of max. capacity estimated by Borg-scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects in permanent atrial fibrillation, willing to participate in a 12 weeks training program and able to give informed consent to participation were eligible for the study.

Exclusion Criteria:

* Subjects with severe refractory hypertension
* previous heart valve surgery, moderate to severe COPD
* restrictive lung disease, moderate to severe asthma
* pregnant or lactating subjects
* patients with a very low life expectancy
* patients who were unable to exercise or comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
cardiac output | participants will be followed for the duration of the intervention, an average of 12 weeks
  participants will be followed for the duration of the intervention, an average of 12 weeks
Quality of life | participants will be followed for the duration of the intervention, an average of 12 weeks
  participants will be followed for the duration of the intervention, an average of 12 weeks
exercise capacity | participants will be followed for the duration of the intervention, an average of 12 weeks
  participants will be followed for the duration of the intervention, an average of 12 weeks

SECONDARY OUTCOMES:
muscle strength | participants will be followed for the duration of the intervention, an average of 12 weeks
  participants will be followed for the duration of the intervention, an average of 12 weeks
biomarkers ANB, BNP | participants will be followed for the duration of the intervention, an average of 12 weeks
  participants will be followed for the duration of the intervention, an average of 12 weeks
Body composition DEXA-scan | participants will be followed for the duration of the intervention, an average of 12 weeks
  participants will be followed for the duration of the intervention, an average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip S Osbak, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Copenhagen, Hvidovre, Denmark